CLINICAL TRIAL: NCT01959321
Title: An Observational Study of Hepatitis C Virus in Pregnancy
Acronym: HCV
Status: Completed | Type: Observational
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: HD36801-HCV; U10HD036801 (NIH); UG1HD087230 (NIH); UG1HD027869 (NIH); UG1HD027915 (NIH); UG1HD034208 (NIH); UG1HD040500 (NIH); UG1HD040485 (NIH); UG1HD053097 (NIH); UG1HD040544 (NIH); UG1HD040545 (NIH); UG1HD040560 (NIH); UG1HD040512 (NIH); UG1HD068282 (NIH); UG1HD068258 (NIH); UG1HD068268 (NIH); UG1HD034116 (NIH); UG1HD087192 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — maternal serum maternal plasma infant serum infant plasma cord blood plasma cord blood buffy coat
Oversight: Data Monitoring Committee: No

SUMMARY:
This multi-center observational study examines risk factors for HCV transmission from mother to baby.

DETAILED DESCRIPTION:
This multi-center observational study examines risk factors for HCV transmission from mother to baby. The study will also assess risk factors associated with Hepatitis C Virus (HCV) infection in pregnant women. Also, the study will describe the outcomes of pregnant women with HCV as well as the outcomes of their infants to 18 months of age.

Approximately 750 HCV antibody positive pregnant women and their infants will be followed from baseline until the infant is 18 months. A randomly selected control cohort of 500 pregnant women who are HCV antibody negative will be followed until delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy
2. An HCV antibody positive screen (case) measured using two FDA-approved ELISA tests, the Abbott Architect version 3.0 system and the Ortho HCV 3.0.
3. Gestational age at screening no later than 23 weeks and 6 days, and gestational age at enrollment no later than 27 weeks and 6 days, based on clinical information and evaluation of the earliest ultrasound as described below.

Exclusion Criteria:

1. Planned termination of pregnancy
2. Known major fetal anomalies or demise
3. Intention of the patient or the managing obstetricians for the delivery to be outside a MFMU Network center, unless special provisions are made to insure infant follow-up at two and 18 months of age.
4. Participation in this study in a previous pregnancy.
5. Unwilling or unable to commit to 18 months of follow-up for HCV positive infants

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with singleton pregnancies presenting for prenatal care prior to 23 weeks, 6 days gestation at Maternal-Fetal Medicine Units (MFMU) Network hospital sites.
Sampling Method: Non-Probability Sample
Enrollment: 772 (Actual)
Dates: Start 2012-10; Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
HCV infection of the offspring | at 2 months and/or 18 months of age
  The primary outcome is HCV infection of the offspring, where infection is defined by satisfying any one of the following criteria:
  * HCV RNA positive (i.e. presence of viral load) by polymerase chain reaction (PCR) test at 2-6 months (2 month visit)
  * HCV RNA positive and HCV antibody positive at the 18-24 months (18 month visit)
  * HCV RNA positive at 18-24 months with a negative HCV antibody at 18-24 months and negative RNA at 2-6 months. However, the positive result must be confirmed by a repeat test on the 18-month sample to qualify.
  * HCV antibody positive at 18-24 months with negative HCV RNA at both visits. However, the positive result must be confirmed by a repeat test on the 18-month sample to qualify.
  * Clinical result that is either HCV RNA positive or HCV antibody positive obtained at 18 months or older with a confirmed clinical diagnosis of HCV, if a central laboratory sample could not be obtained at 18-24 months.

SECONDARY OUTCOMES:
Gestational age at delivery | at birth
Preterm delivery < 37 weeks of gestation | at birth
Gestational diabetes mellitus (GDM) | during pregnancy
Vaginal bleeding during pregnancy | during pregnancy
Preeclampsia | during pregnancy
Cholestasis | during pregnancy
Viral load in infant | at birth, 2 months, and 18 months
HCV antibody status in infant | at 18 months of age
  positive or negative
Birth weight of infant | at birth
Hyperbilirubinemia | at birth
  Peak total bilirubin of at least 15 mg% or the use of phototherapy
Neonatal intensive care unit (NICU) admission | at birth
Small for gestational age | at birth
  Defined as less than the 5th percentile birth weight for gestational age at birth, assessed specifically by sex and race of the infant based on United States birth certificate data
Neonatal infections | at birth
  sepsis and pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Monica Longo, M.D., Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Rebecca Clifton, PhD, Principal Investigator — The George Washington University Biostatistics Center; Mona Prasad, DO, MPH, Study Chair — Ohio State University
Locations (17):
- United States (17):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Stanford University, Stanford, California
  - University of Colorado, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas - Galveston, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be shared per NIH policy after the completion and publication of the main analyses.

REFERENCES:
- [Derived] Grasch JL, de Voest JA, Saade GR, Hughes BL, Reddy UM, Costantine MM, Chien EK, Tita ATN, Thorp JM Jr, Metz TD, Wapner RJ, Sabharwal V, Simhan HN, Swamy GK, Heyborne KD, Sibai BM, Grobman WA, El-Sayed YY, Casey BM, Parry S; for the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network*. Breastfeeding Initiation, Duration, and Associated Factors Among People With Hepatitis C Virus Infection. Obstet Gynecol. 2024 Mar 1;143(3):449-455. doi: 10.1097/AOG.0000000000005499. Epub 2024 Jan 4. PMID 38176013
- [Derived] Prasad M, Saade GR, Sandoval G, Hughes BL, Reddy UM, Mele L, Salazar A, Varner MW, Gyamfi-Bannerman C, Thorp JM Jr, Tita ATN, Swamy GK, Chien EK, Casey BM, Peaceman AM, El-Sayed YY, Iams JD, Gibbs RS, Sibai B, Wiese N, Kamili S, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Hepatitis C Virus Antibody Screening in a Cohort of Pregnant Women: Identifying Seroprevalence and Risk Factors. Obstet Gynecol. 2020 Apr;135(4):778-788. doi: 10.1097/AOG.0000000000003754. PMID 32168224